CLINICAL TRIAL: NCT03024320
Title: Scale Up Evaluation of a Physical Activity Program for Adults With Physical Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other); Tanner Foundation for Multiple Sclerosis (Other)
Responsible Party: Principal Investigator, James Rimmer, Professor and Director of UAB/Lakeshore Collaborative, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: F160923002
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Physical Disability

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with three arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- M2M (Experimental): A theory-driven eHealth platform and innovative physical activity program referred to as movement-to-music (M2M), delivered customized and for the home-based for adults with physical disability.
  Interventions: Behavioral: M2M
- M2Mplus (Experimental): A theory-driven eHealth platform and innovative physical activity program referred to as movement-to-music (M2M), delivered customized and for the home-based for adults with physical disability. This arm also includes a social networking platform where participants will be able to interact and encourage one another through the program, as well as group-based tele-coaching session.
  Interventions: Behavioral: M2M
- Attention Control (Active Comparator): Participants receive health-focused articles and infographics throughout 48 weeks and receive a Fitbit.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: M2M — An eHealth platform has been designed to deliver a home-based package using the extensive set of movement patterns that have been adapted for people with a range of physical/mobility disability, called Movement-To-Music (M2M). The M2M prescription will be based on the participant's baseline level of health, function and fitness. Each movement pattern will be available in three different positions - standing, standing with support (chair) and seated. The duration of each M2M session will be gradually increased during the Adoption phase from three 20-minute sessions (10 min. aerobic & 10 min. strength) during weeks 1 to 3 (60 min/wk), to 45-min sessions (30 min. aerobic & 15 min. strength) during weeks 4 to 6 (135 min/wk), and to 50-min sessions (150 min/week) during weeks 7 to 12 (excluding 5-min warmup and 5-min cool down).
  Arms: M2M; M2Mplus
Behavioral: Attention Control — Telecoaching on health-based topics, not including physical activity.
  Arms: Attention Control

SUMMARY:
The study uses a theory-driven eHealth platform and innovative physical activity (PA) program referred to as movement-to-music (M2M) to deliver a customized, home-based PA intervention for adults with physical disability (PWD). Participants will be recruited through a large physical medicine and rehabilitation network of clinics specializing in treating patients with physical disability. Participants will be randomized to one of three groups: a) M2M; b) M2M plus social networking (M2Mplus); and c) attention control (AC). Participants will be followed for 48 weeks to obtain objective measures on physical activity, fitness and self-reported measures on health at four time points. The study will compare the effectiveness of M2M and M2Mplus in increasing physical activity and adherence compared to the AC group, estimate the improvements in health of M2M and M2Mplus compared to the AC group, and examine the mediators and moderators of the hypothesized treatment effect to understand for whom and how the intervention is effective. This multi-level, scalability study will strengthen our understanding of the potential benefits of eHealth to eliminate barriers to PA participation among PWD.

DETAILED DESCRIPTION:
This study contains two intervention groups and one attention control group. Participation by each individual will include recruitment, screening, consent, baseline assessment, randomization to one of the three groups, adoption and transition phase assessments and post-assessment. The intervention will be delivered in three phases: (1) Adoption (weeks 1 to 12); (2) Transition (weeks 13 to 24); and (3) Maintenance (weeks 25 to 48). This phased approach will allow us to gradually adjust the dosage of the intervention and be able to capture the effects of the change in dosage. The study includes an eHealth platform to deliver M2M content (for the M2M and M2Mplus groups).

ALL GROUPS (attention control, M2M, M2Mplus) All groups will be involved in baseline, 3-month, and post-testing, which is being conducted at Lakeshore Foundation and Tanner Foundation for Multiple Sclerosis. In response to limited business operations, there is now an option for enrolling virtually by completing tele-assessments, which are completed through Zoom. All study measures are completed using the tele-assessment with the exception of a sub-max arm ergometer test. These assessments include short forms (SFs) developed by the National Institutes of Health (NIH) Patient-Reported Outcome Measurement Information System (PROMIS) which will be used to measure symptoms and quality of life indicators. Cardiorespiratory endurance will be measured by a sub-max arm ergometer test while strength is measured by a grip strength dynamometer. Anthropometrics assessments include height, weight, BMI and waist circumference. Other assessments include social support, self-efficacy, self-regulation, outcome expectancies, barriers, physical function, and blood pressure. Copies of all assessment forms, surveys, and procedures are attached to this protocol.

Physical activity and adherence are the key outcome measures. Physical activity will be estimated by the self-reported Godin Leisure Time Exercise Questionnaire (GTLEQ) and monitored for implementation by a Fitbit activity monitor. FitBit HR 2 (the most popular version of commercial accelerometers) will be given to all study participants to track their rate of physical activity. Fitbit trackers use a 3-axis accelerometer to capture motions, making its activity measurements more precise than older, single-axis pedometers, which enable us to measure physical activity adherence in PWD. The data, including personal health information (PHI) such as date of birth, height and weight needed for Fitbit setup,are uploaded to a protected server run by FitBit. This happens automatically and does not require any type of manual setup by the participant. The uploaded data will only contain the sensor's unique identification code and no personally identifiable information. The project's eHealth platform will connect to the FitBit servers through an application program interface, to locally host the data for further analysis. The project coordinator will have access to participants' activity data through their respective dashboards on the eHealth platform. The activity data, coupled with our advanced eHealth tracking routines, will enable the statistician to match the minutes of videos watched (dosage) and the change in physical activity (from FitBit steps). Participants will wear the FitBit accelerometer at all times so that the investigators can also track any changes in PA across a 24-hr period. To monitor and ensure that the FitBit sensor is worn, a monitoring system will be included that will send an automated text message or voicemail when a participant fails to wear the FitBit for more than 12 hours. Adherence rate of a participant is defined as the percentage of 48 weeks a participant meets the study protocol's physical activity target. This will enable a comparable measure of adherence across the intervention and control arms.

M2M/M2Mplus GROUPS Participants in the M2M and M2Mplus group receive the telehealth exercise training program. Our advanced eHealth platform designed for the National Center on Health, Physical Activity and Disability's (NCHPAD) 14-Weeks To a Healthier You program includes the foundational elements required for rapid deployment of the M2M content. The onsite M2M program currently at Lakeshore Foundation has been converted into a home-based package using extensive sets of movement routines that have been adapted for people with a range of physical/mobility disability. The M2M movement routines and the positions used to perform the movement routines are prescribed based on participants' physical function. Each movement routine will be available in different choices of music type- to enable participants exercise with the music type they prefer.

The M2M exercise videos are created to incorporate a holistic movement routine. Each exercise video includes five components: warm-up/range of motion exercise, strength exercise, aerobic exercise, functional strength/balance exercise, and cool-down/breathing. The movements are choreographed and adapted to target these components by experienced dance instructors. Exercise equipment, such as TheraBand or hand weights, can be used but is not required. All M2M movement routines will be reviewed by a physical therapist/exercise physiology co-investigator (Brown) for clarity and safety. The duration and movement complexity of each M2M session will be gradually increased from 30-minute sessions (5-min range of motion movement routine, 10-min strength movement routine, 10-min aerobic movement routine, 5-min cool down/breathing) to 60-min sessions (5-min range of motion movement routine, 10-min strength movement routine, 30-min aerobic movement routine, 10-min functional strength/balance routine, and 5-min cool down/breathing) throughout the Adoption and Transition phases of the intervention. The duration and movement complexity of the M2M sessions will be kept consistent during the maintenance phase (5-min range of motion movement routine, 10-min strength movement routine, 30-min aerobic movement routine, 10-min functional strength/balance routine, and 5-min cool down/breathing). Participants will be encouraged to work at their self-selected pace and comfort level, meaning that they can pause the M2M video anytime when they need a break and resume when they are ready. Participants do not have to complete the entire 50 minutes if they do not feel comfortable in doing so. Participants will provide feedback on a brief electronic form uploaded to the project coordinator on how they performed each set of M2M movement routines and what they liked/disliked about the movement routines, preferably within two hours after completing a M2M session.

Each M2M session will start with brief exercise reminders such as maintaining good form or using the 'talk test' to ensure that the intensity level is not outside the individual's comfort level. The participant can stop the video to rest at any time by touching their tablet/electronic device and then returning to the same segment so that 'dosing' remains consistent across all participants, albeit some participants who are less fit may need longer and more frequent rest intervals during the first few weeks of training. The eHealth platform will be password protected to enable detailed usage tracking. The M2M videos will be offered through a YouTube playlist player, which offers a seamless experience and can quickly be played and paused with a minimum number of clicks. To monitor the delivery of the videos, event tracking will be used. This will help the researchers know precisely which of the videos were viewed and for how long.

At week 5 of the exercise program, individuals who are not engaging in exercise by using their Fitbit or clicking on videos, they will be contacted by research staff for a brief interview. The purpose of this interview is to understand lack of participation in the exercise intervention and perhaps re-engage the participant. At week 12 of the exercise program, individuals who are not engaging in exercise since week 5 by using their Fitbit or clicking on videos, they will be contacted by research staff for a brief interview. No identifiable information will be link the interview to the participant.

M2Mplus GROUP ONLY For the M2Mplus group, a social networking system (SNS) is integrated into the eHealth platform. SNS features allows users to engage in conversation and other forms of social interactions (such as posting a rating score on a certain video or movement sequence they liked or disliked) across the eHealth platform. The participant's physician or designated nurse will also have access to the SNS to build a close asynchronous relationship with their patient. The social networking component of the platform includes all essential building blocks of social media including (1) identity; (2) sharing; (3) presence; (4) relationships; (5) reputations; (6) groups, and; (7) conversations,105 and will be repurposed and enhanced from the SNS developed for the NCHPAD 14 Weeks To A Healthier You online program, where users expressed a strong desire to be able to closely interact with fellow participants (see sample quote in box to the right). The SNS features of the intervention are developed using the popular open source SNS framework "Elgg." Additionally, participants in the M2Mplus group receives a group-basedcoaching session led by the research team who has expertise in motivational interviewing strategies. The coaching sessions will follow the framework developed by our consultant exercise psychologist and used in our previous research with adults with physical disability. The calls will focus on the topics related to social support, overcoming barriers, and preventing relapse. These sessions will be held weekly during the Adoption phase (weeks 1-12), biweekly during the Transition phase (weeks 13-24), and monthly during the Maintenance phase (weeks 25-48).

ELIGIBILITY:
Inclusion Criteria:

* Underactive adults (< 60 minutes of moderate intensity exercise per week in the last month)
* Diagnosis of a physical/mobility disability by their physician
* Working age adult 18 to 70 yrs. of age
* No physician contraindications to exercise and written physician approval to participate in the study
* Not currently enrolled in a structured exercise program over the past 6 months
* Have the ability to use upper, lower or both sets of extremities to exercise
* Must have the ability to converse and read English

Exclusion Criteria:

* Medically unstable to perform home exercise as determined by their physician
* High level tetraplegia and unable to use arms or legs to exercise
* Cognitive impairment that may preclude self-directed daily activities
* No internet access.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 48 weeks
  Godin Leisure Time Exercise Questionnaire (GLTEQ) provides the Health Contribution Score which is calculated based on the number of minutes of physical activity multiplied by intensity level.
Completing program content | 48 weeks
  Tracking tablet and Fitbit activity to know if participants are watching the exercise videos.

SECONDARY OUTCOMES:
Cardiorespiratory Endurance | baseline, 12 weeks, 48 weeks
  Sub-max Arm Ergometer Test
Strength | baseline, 12 weeks, 48 weeks
  grip strength
Physical Function | baseline, 12 weeks, 48 weeks
  physical performance battery
Blood pressure | baseline, 12 weeks, 48 weeks
  Two readings prior to exercise using BP cuffs.
Height | baseline, 12 weeks, 48 weeks
  Standing or lying measured in inches and centimeters.
Weight | baseline, 12 weeks, 48 weeks
  Scale
BMI | baseline, 12 weeks, 48 weeks
  Body Mass Index
Waist Circumference | baseline, 12 weeks, 48 weeks
  Hip and naval.
Barriers to Physical Activity and Disability Survey | baseline, 12 weeks, 24 weeks, 48 weeks
  Barriers to Physical Activity for people with disabilities.
Outcome Expectations for Exercise Scale | baseline, 12 weeks, 24 weeks, 48 weeks
  Survey of social cognitive theory construct.
Strategies for Physical Activity Scale | baseline, 12 weeks, 24 weeks, 48 weeks
  Self-regulation measurement.
Physical Activity Self-efficacy Scale | baseline, 12 weeks, 24 weeks, 48 weeks
  Survey of social cognitive theory construct.
Demographics | baseline
  questionnaire
Physical Functioning | baseline, 12 weeks, 24 weeks, 48 weeks
  NIH PROMIS
Sleep | baseline, 12 weeks, 24 weeks, 48 weeks
  Secondary health conditions NIH PROMIS
Fatigue | baseline, 12 weeks, 24 weeks, 48 weeks
  NIH PROMIS
Pain Intensity | baseline, 12 weeks, 24 weeks, 48 weeks
  Secondary health conditions NIH PROMIS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai BW, Rimmer JH, Yates A, Jeter A, Young HJ, Thirumalai M, Mehta T, Wilroy J. Critical factors influencing the decision to enroll in a physical activity intervention among a predominant group of adults with spinal cord injury: a grounded theory study. Spinal Cord. 2021 Jan;59(1):17-25. doi: 10.1038/s41393-020-0530-7. Epub 2020 Aug 3. PMID 32747672
- [Background] Rimmer JH, Mehta T, Wilroy J, Lai B, Young HJ, Kim Y, Pekmezi D, Thirumalai M. Rationale and design of a Scale-Up Project Evaluating Responsiveness to Home Exercise And Lifestyle Tele-Health (SUPER-HEALTH) in people with physical/mobility disabilities: a type 1 hybrid design effectiveness trial. BMJ Open. 2019 Mar 30;9(3):e023538. doi: 10.1136/bmjopen-2018-023538. PMID 30928927
- [Background] Lai B, Wilroy J, Young HJ, Howell J, Rimmer JH, Mehta T, Thirumalai M. A Mobile App to Promote Adapted Exercise and Social Networking for People With Physical Disabilities: Usability Study. JMIR Form Res. 2019 Mar 19;3(1):e11689. doi: 10.2196/11689. PMID 30888325
- [Background] Wilroy JD, Lai B, Davlyatov G, Mehta T, Thirumalai M, Rimmer JH. Correlates of adherence in a home-based, self-managed exercise program tailored to wheelchair users with spinal cord injury. Spinal Cord. 2021 Jan;59(1):55-62. doi: 10.1038/s41393-020-0497-4. Epub 2020 Jun 15. PMID 32541883
- [Background] Wilroy J, Lai B, Currie M, Young HJ, Thirumalai M, Mehta T, Giannone J, Rimmer J. Teleassessments for Enrollment of Adults With Physical or Mobility Disability in a Home-Based Exercise Trial in Response to COVID-19: Usability Study. JMIR Form Res. 2021 Nov 18;5(11):e29799. doi: 10.2196/29799. PMID 34792477
- See also: Study Website — http://superhealthstudy.org